CLINICAL TRIAL: NCT06767046
Title: An Exploratory Study to Evaluate the Safety and Preliminary Efficacy of KRAS-Specific Autologous TCR-T Cells in Advanced Solid Tumors
Brief Title: KRAS-Specific Autologous TCR-T Cell Therapy for KRAS Mutation in Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Corregene Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTKVA11-2311C
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Colorectal; Pancreatic; Non-small Cell Lung Cancer (NSCLC)
Keywords: KRAS G12V; immunotherapy; T cell; Adoptive cell therapy; T cell receptor; TCR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KRAS-specific Autologous TCR-T cell injection (Experimental): KRAS-specific Autologous TCR-T cell injection (5×10⁹, 1×10¹°, or 2×10¹° TCR-T cells per dose) with preconditioning lymphodepletion using Fludarabine and Cyclophosphamide, followed by IL-2 support
  Interventions: Drug: KRAS-specific Autologous TCR-T cell injection

INTERVENTIONS:
Drug: KRAS-specific Autologous TCR-T cell injection — Drug1 : Fludarabine + Cyclophosphamide Drug2 :Interleukin 2 Drug3 :KRAS-specific Autologous TCR-T cell injection
  Other Names: CRTKVA11-N04

SUMMARY:
This is a single-center, open-label, single-arm, dose-escalation study aimed at evaluating the safety and preliminary efficacy of KRAS-specific autologous TCR-T cells in patients with advanced solid tumors harboring KRAS G12V mutation.

DETAILED DESCRIPTION:
T cell receptor-gene engineered T cells (TCR-T) therapy is a highly targeted form of cellular immunotherapy. It is safer than Chimeric Antigen Receptor T-Cell Immunotherapy (CAR-T) and is currently a hot topic in immunotherapy. In the case of advanced pancreatic cancer with KRAS mutations, the infusion of TCR-T cells has achieved good efficacy and safety, further suggesting the promising prospects of TCR-T cell immunotherapy for advanced solid tumors with KRAS G12V mutation.

It is planned to enroll 9 - 18 patients with advanced solid tumors who have KRAS G12V mutation and HLA-A*11:01 genotype, and have failed standard treatments. A single-center, open-label, single-arm study design will be adopted. The KRAS-specific autologous TCR-T cell injection will be used to treat these patients. The primary endpoint is safety, and the secondary endpoints include efficacy, cell activity, etc. It is planned to select three dose groups with 5×10⁹, 1×10¹⁰, and 2×10¹⁰ TCR-T cells respectively, and conduct dose escalation using a 3 + 3 study design.

The key steps involved in the study are the preparation and quality control of TCR-T cells, lymphocyte depletion (lymphodepletion), and the infusion of autologous TCR-T cell injection. Record and promptly handle specific adverse reactions of cellular immunotherapy, such as cytokine release syndrome (CRS), various other adverse events, off-target effects of TCR-T, and adverse events related to tumorigenic potential, etc., to obtain safety data. It is hoped that the results of this study will bring a new future for patients with advanced solid tumors with specific KRAS mutations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years.
* Histologically or cytologically confirmed advanced solid tumors (e.g., colorectal cancer, pancreatic cancer, NSCLC) with KRAS G12V mutations and HLA-A*11:01 genotype.
* Failed standard therapies or no effective treatment available.
* ECOG performance status of 0-1.
* Life expectancy of ≥3 months.
* Presence of at least one measurable lesion as defined by RECIST 1.1 criteria.
* Female patients of childbearing potential must agree to use highly effective contraceptive methods during the study and for at least 6 months after the last dose. A negative pregnancy test within 7 days prior to treatment initiation is required.
* Written informed consent provided by the patient, with an expectation of compliance with study procedures.

Exclusion Criteria:

* 1.Prior treatment with gene-modified T-cell therapies.
* Current treatment with T-cell suppressive agents (e.g., cyclophosphamide, FK506, tripterygium glycosides) or T-cell stimulants.
* Chemotherapy, targeted therapy, immunotherapy, or investigational drugs administered within 2 weeks, or radiotherapy within 4 weeks prior to enrollment.
* Significant organ dysfunction, as evidenced by:

  * leukocytes<3.0 x 109/L
  * absolute neutrophil count >1.5 x 109/L
  * hemoglobin<90g/L
  * platelets <100 x 109/L
  * Creatinine>1.5×ULN or creatinine clearance <50mL/min
  * lymphocytes<0.5 x 109/L
  * total bilirubin>3×ULN; ALT/AST>3×ULN (or >5× ULN in patients with liver metastases)
  * INR/APTT>1.5×ULN；
  * SpO2≤93%
* Presence of serious diseases and comorbidities, including but not limited to: severe heart disease, cerebrovascular disease, seizures, poorly controlled diabetes (such as Type 1 diabetes or insulin-dependent diabetes), pancreatic dysfunction, severe infections, active gastrointestinal ulcers, gastrointestinal bleeding, mechanical or paralytic bowel obstruction, pulmonary fibrosis, renal failure, respiratory failure, etc.
* History of severe cardiovascular diseases within the past 6 months, including but not limited to: myocardial infarction, severe or unstable angina, coronary artery or peripheral artery bypass surgery, New York Heart Association (NYHA) Class III or IV heart failure, etc.
* Left ventricular ejection fraction (LVEF) < 50%.
* Symptomatic brain metastases unless stabilized with prior treatment (e.g., surgery or radiotherapy).
* Known history of myelodysplastic syndrome, lymphoma, or other malignancies.
* Known allergy to albumin, investigational drugs, or their excipients.
* Active autoimmune diseases, including but not limited to acquired/congenital immunodeficiency, organ transplantation, autoimmune hepatitis, systemic lupus erythematosus, or inflammatory bowel disease.
* Active hepatitis B, hepatitis C, or HIV infection.
* Pregnancy or breastfeeding.
* Uncontrolled mental or neurological disorders.
* Any condition deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2025-02-18 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related AEs, AEs of special interest and serious adverse events (SAEs) | 2 years
  Incidence of treatment related AEs, AEs of special interest and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  Assessed by RECIST 1.1
Disease Control Rate (DCR) | 2 years
  Assessed by RECIST 1.1
Duration of Response (DOR) | 2 years
  Assessed by RECIST 1.1
Progression-Free Survival (PFS) | 2 years
  Assessed by RECIST 1.1
Overall Survival (OS) | 2 years
  Overall survival was defined as the time from KRAS-Specific Autologous TCR-T Cell infusion to the date of death

CONTACTS AND LOCATIONS:
Locations (1):
- Captital Medical University Affiliated Beijing Ditan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No